CLINICAL TRIAL: NCT06935045
Title: Evaluating How Alcohol Impacts Physiological Responses and Perception During Heat Exposure
Brief Title: Ethanol Consumption in the Heat
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lakehead University (Other)
Responsible Party: Principal Investigator, Nicholas Ravanelli, Assistant Professor, Lakehead University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1469888
Record Dates: First submitted 2025-04-01; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Consumption; Heat Stress; Age
Keywords: alcohol; heat stress; heat wave; sweating; core temperature; micturition; perception; behaviour
MeSH Terms: conditions — Alcohol Drinking; Heat Stress Disorders; Behavior | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (non-alcoholic beverage)
  Interventions: Drug: Placebo Beverage
- Alcohol (Active Comparator): Consumption of alcohol beverages: females 0.75 ± 0.1 grams of ethanol/kilogram body mass; males 1.0 ± 0.1 grams of ethanol/kilogram body mass
  Interventions: Drug: Alcohol (Ethanol)

INTERVENTIONS:
Drug: Placebo Beverage — Participants rest in a climate controlled room maintained at 40°C and 30%RH for 120 minutes follow placebo beverage consumption (180 minutes total).
  Arms: Placebo
Drug: Alcohol (Ethanol) — Participants rest in a climate controlled room maintained at 40°C and 30%RH for 120 minutes follow alcoholic beverage consumption (180 minutes total).
  Arms: Alcohol

SUMMARY:
Climate change has significantly increased the earth's average surface temperature and heat waves have been predicted to increase in frequency, intensity and duration. Extreme heat events have increased the susceptibility to heat-related illnesses, such as heat exhaustion, heat stroke or death. Heat health action plans have been designed to advertise cooling behaviours to mitigate physiological strain. Heat health action plans suggest avoiding alcohol consumption during extreme heat as it may increase dehydration and impair behavioural or physiological temperature regulation and thermal perception. Regardless of these messages, alcohol sales continue to remain high during the summer months year after year, and 1/5 of adults identify alcohol as a hydration strategy during extreme heat events. A recent scoping review investigating the effects of alcohol and heat has demonstrated that acute alcohol consumption does not negatively influence thermoregulation, hydration, or hormone markers of fluid balance in the heat compared to a control fluid (https://doi.org/10.1186/s12940-024-01113-y). Further, alcohol consumption may elicit sex- and age-specific alterations in physiological and perceptual responses, neither of which have been explored.

Therefore, this study aims to comprehensively evaluate how alcohol consumption systematically alters physiological responses and perceptions during conditions similar to those experienced indoors during extreme heat events in younger and older adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female above the age of 19
* Able to provide informed consent

Exclusion Criteria:

* History of cardiovascular disease, cancer, type 1 or 2 diabetes, chronic obstructive pulmonary disorder, cystic fibrosis, or alcohol addiction or dependence
* Been hospitalized due to COVID-19
* Pregnant/Breastfeeding
* Scoring an eight or above on the Alcohol Use Disorders Identification Test (AUDIT)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | measured at baseline (pre drink), and every 30 minutes following consumption (up to 120 minutes).
  3-lead electrocardiogram
Skin Temperature | measured at baseline (pre drink), and every 30 minutes following consumption (up to 120 minutes).
  Mean skin (4 sites)
Core Temperature | measured at baseline (pre drink), and every 30 minutes following consumption (up to 120 minutes).
  measured rectally
Blood Pressure | measured at baseline (pre drink), and every 30 minutes following consumption (up to 120 minutes).
  ECG-gated blood pressure cuff
Heart Rate Variability | measured at baseline (pre drink), and every 30 minutes following consumption (up to 120 minutes).
Arrythmia presence | measured at baseline (pre drink), and every 30 minutes following consumption (up to 120 minutes).
Whole-body Sweat Loss | mass measured at baseline and end heat stress.
  Difference in mass from baseline to end heat stress
Postural Sway via the Romberg Test | measured at baseline (pre drink), and every 30 minutes following consumption (up to 120 minutes).
  The total movement of the body around the center of mass with feet together
Skin Blood Flow | measured at baseline (pre drink), and every 30 minutes following consumption (up to 120 minutes).
Urine Output | Total urine output (e.g. volume) from baseline to immediately following 120 minutes of heat stress
ASHRAE seven-point thermal sensation scale | measured at baseline (pre drink), and every 30 minutes following consumption (up to 120 minutes).
5-Point Thermal Comfort Scale | measured at baseline (pre drink), and every 30 minutes following consumption (up to 120 minutes).
  Thermal comfort scale with 1- comfortable and 5 - very uncomfortable

SECONDARY OUTCOMES:
Subjective Blood Alcohol Concentration (visual analog scale 0.0 - 0.20) | measured at baseline (pre drink), and every 30 minutes following consumption (up to 120 minutes).
  Visual analog scale with left and right anchors of 0.0 and 0.20, respectively, with markers every 0.005 increment
Blood Alcohol Concentration | measured at baseline (pre drink), and every 30 minutes following consumption (up to 120 minutes).
  Measured using a police grade portable breathalyzer

CONTACTS AND LOCATIONS:
Locations (1):
- Lakehead University, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared on the Open Science Framework following publication of results
Access Criteria: Anyone will have access

REFERENCES:
- [Background] Morris NB, Ravanelli N, Chaseling GK. The effect of alcohol consumption on human physiological and perceptual responses to heat stress: a systematic scoping review. Environ Health. 2024 Sep 12;23(1):73. doi: 10.1186/s12940-024-01113-y. PMID 39267036